CLINICAL TRIAL: NCT04891315
Title: Measuring Soluble Vascular Adhesion Protein-1 as a Potential Biomarker for Predicting Pregnancy Problems
Brief Title: Measuring sVAP-1 as a Predictor of Pregnancy Problems
Status: Terminated | Type: Observational
Why Stopped: A recalculation of sample size following preliminary results showed that the study was not feasible due to the requirement of a much larger sample size to reach significance. This would not be possible without significant additional funding.
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0820; 289532 (Other: IRAS); 21/EM/0090 (Other: Leicester Central Research Ethics Committee)
Record Dates: First submitted 2021-04-26; First posted 2021-05-18 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-09

CONDITIONS: Pregnancy Complications
Keywords: Hypertension in pregnancy; Pre-eclampsia; Gestational diabetes; Fetal growth restriction; Large for gestational age; Stillbirth; Miscarriage
MeSH Terms: conditions — Pregnancy Complications; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Diabetes, Gestational; Fetal Growth Retardation; Stillbirth; Abortion, Spontaneous | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Women aged 16+ in early pregnancy (before 20 weeks of gestation).
  Interventions: Diagnostic Test: Blood test for soluble VAP-1 (sVAP-1).

INTERVENTIONS:
Diagnostic Test: Blood test for soluble VAP-1 (sVAP-1). — ~5ml blood will be taken and sVAP-1 will be measure by Enzyme linked Immunosorbent Assay

SUMMARY:
Pre-eclampsia is a common pregnancy disorder defined as high blood pressure and protein in the urine after 20 weeks of pregnancy. It affects the function of the placenta and can cause severe complications, e.g, stroke, multiple organ damage and seizures for the mother, and fetal growth restriction or stillbirth for the baby. Pre-eclampsia can also cause long term health problems for mother and baby.

Currently, there is no test that can predict whether someone will develop pre-eclampsia, so nothing is done to intervene before the problems begin.

Results from their previous work suggest that the investigators may have found something that can be measured in a blood sample that can predict which women might develop pre-eclampsia. It is a protein known as Vascular Adhesion Protein-1 (VAP-1), and our evidence points at it being involved in the embryo attaching to the womb and also in helping the development of the placenta by helping to get the right cells to where they are needed.

The investigators will test blood samples from 451 pregnant women who come to the Leicester Royal Infirmary for routine bloods and their first pregnancy dating scan. The investigators will then follow the outcomes of the pregnancy to see if VAP-1 in the blood of women who develop pre-eclampsia (or other pregnancy complications) is different from the ones who do not develop pregnancy complications. The ability to predict women at higher risk of pregnancy complications would ensure the application of timely interventions and appropriate management of the conditions that may help to prevent complications both during pregnancy and later life.

The study is expected to last approximately 30 weeks and the participants will be asked to give one extra tube of blood whilst having their routine bloods taken and to also consent to follow up of medical records until the end of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are in early pregnancy (<20 weeks gestational age).
* 16 years and above
* Patient consents to take part in the study

Exclusion Criteria:

* Patient declines to be involved in the study
* Unsuccessful venepuncture

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — No: Eligibility is not based on gender
Study Population: All patients being given an appointment for a routine dating scan and blood test at the Leicester Royal Infirmary will have a copy of the patient information sheet included within their appointment letter and will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Correlation of sVAP-1 levels with pregnancy complications: Pre-eclampsia | During pregnancy up to 42 weeks
  Diagnosis of pre-eclampsia defined as:
  New-onset hypertension (>140 mm Hg systolic or >90 mm Hg diastolic) after 20 weeks of pregnancy and the coexistence of one or both of the following new-onset conditions:
  Proteinuria (urine protein:creatinine ratio ≥30 mg/mmol, or albumin:creatinine ratio ≥8 mg/mmol, or ≥1 g/L [2+] on dipstick testing) Other maternal organ dysfunction.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with pregnancy complications: hypertension in pregnancy | During pregnancy up to 42 weeks
  Diagnosis of hypertension in pregnancy defined as:
  Systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mmHg.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with pregnancy complications: Gestational diabetes. | During pregnancy up to 42 weeks
  Diagnosis of gestational diabetes defined as:
  A fasting plasma glucose level of 5.6 mmol/litre or above or A 2-hour plasma glucose level of 7.8 mmol/litre or above
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with Fetal outcomes: Stillbirth | During pregnancy from 24 to 42 weeks
  Stillbirths will be defined as:
  The death of a baby before or during birth after 24 weeks of gestation.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with Fetal outcomes: Fetal growth restriction | During pregnancy up to 42 weeks
  Fetal growth restriction will be defined as:
  Estimated fetal weight >10th centile for gestational age.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with Fetal outcomes: Fetal macrosomia | During pregnancy up to 42 weeks
  Fetal macrosomia,will be defined as:
  Estimated fetal weight >90th centile for gestational age.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with Fetal outcomes: Preterm labour | During pregnancy up to 37 weeks
  Preterm labour be defined as:
  Birth <37 weeks.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with Fetal outcomes: Miscarriage | During pregnancy up to 24 weeks
  Miscarriage will be defined as:
  Occurrence of spontaneous abortion <24 weeks' gestation.
  sVAP-1 levels will be measured by ELISA

SECONDARY OUTCOMES:
Correlation of sVAP-1 levels with patient characteristics: Age | At time of recruitment
  Age will be measured in years.
  sVAP-1 levels will be measured by ELISA
Correlation of sVAP-1 levels with patient characteristics: Weight | During pregnancy up to 42 weeks
  Weight will be measured in kilograms.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: BMI | During pregnancy up to 42 weeks
  Weight and height will be combined to report BMI in kg/m^2.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Ethnicity | At time of recruitment
  Ethnicity will be recorded as described on the medical records of the patient.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Smoking status | During pregnancy up to 42 weeks
  Smoking status will be recorded as current/ex/never.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Gestation at time of recruitment | At time of recruitment
  Gestation at time of recruitment will be measured in weeks.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Parity | At time of recruitment
  Parity will be recorded as the number of births with a gestational age of 24 weeks.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Gravidity | At time of recruitment
  Gravidity will be recorded as the total number of pregnancies.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Pre-existing medical conditions | At time of recruitment
  Pre-existing medical conditions will be recorded as reported on the patient's medical records.
  sVAP-1 levels will be measured by ELISA.
Correlation of sVAP-1 levels with patient characteristics: Medications at time of booking | At time of recruitment
  Medications at time of booking will be recorded as reported on the patient's medical records.
  sVAP-1 levels will be measured by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester Royal Infirmary, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data.